CLINICAL TRIAL: NCT05927870
Title: Ultrasound Guided Percutaneous Cholecystostomy as Preoperative Step for Obstructive Gallbladder Diseases.
Brief Title: Ultrasound Guided Percutaneous Cholecystostomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basma Fawzy Abd Elhameed Ali, Resident doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: percutaneous cholecystostomy
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Gall Bladder Disease
MeSH Terms: conditions — Gallbladder Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyocele (Experimental): obstructed gallbladder with infection on top
  Interventions: Procedure: pigtail

INTERVENTIONS:
Procedure: pigtail — placing a small amount of local anaesthetic subcutaneously at the site of the gallbladder, a skin incision was made through which the catheter was introduced. A 7-Fr pigtail catheter was used in all cases . If possible, the catheter was introduced into the gallbladder after passing through the liver. The catheter was thereafter fixed, either by an internal locking device or by means of a suture to the skin. The catheter was rinsed with saline solution daily in order to prevent clogging.

SUMMARY:
Surgical cholecystostomy has proven value in the management of both inflammatory and obstructive biliary tract disease

DETAILED DESCRIPTION:
The etiology of biliary obstruction can be benign or malignant. Benign disease, such as calculi, strictures, or pancreatitis, can be common causes in adult patients [5], whereas benign strictures including posttransplant anastomotic strictures and strictures secondary to hepatic artery insufficiency, stone disease, infection, and iatrogenic causes can be seen in children [6]. Obstruction can also be seen in the setting of biliary tract abnormalities, such as biliary atresia in neonates and symptomatic choledochal cysts, autoimmune pancreatitis, and sclerosing cholangitis in older children [7]. Biliary obstruction secondary to neoplasm commonly occurs with pancreatic cancer, cholangiocarcinoma, or metastases in adult patients and biliary rhabdomyosarcoma or neuroblastoma in younger patients [8].

The question remains as to whether all patients undergoing PCT drainage require a definitive cholecystectomy. Previous publications have suggested that there is a reluctance to use PCT in older and comorbid patients due to concerns of potentially committing such patients to an interval surgical procedure for which they may not be suitable.

ELIGIBILITY:
Inclusion Criteria:

* Pyocele of the gallbladder
* Mucocele of the gallbladder
* Perforated gallbladder
* Malignant causes of gallbladder obstruction

Exclusion Criteria:

* Uncontrolled bleeding disorders

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
value of cholecystostomy as preoperative step in critically ill patients | basline
  The aim of this study was to assess the clinical outcomes of PCT use, with particular emphasis on a subgroup of patients who did not proceed to cholecystectomy.

REFERENCES:
- [Background] Akhan O, Akinci D, Ozmen MN. Percutaneous cholecystostomy. Eur J Radiol. 2002 Sep;43(3):229-36. doi: 10.1016/s0720-048x(02)00158-4. PMID 12204405
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12204405/